CLINICAL TRIAL: NCT05984459
Title: Type 2 Diabetes Treatment and Remission With a Very Low-Calorie Ketogenic Diet (VLCKD) and Lifestyle Changes
Status: Completed | Type: Observational
Sponsor: Cabinet Medical (Other)
Collaborators: Trialance SCCL (Industry)
Responsible Party: Sponsor
Other Study IDs: FMH Endocrinol and Diabetol
Record Dates: First submitted 2023-07-24; First posted 2023-08-09 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-08

CONDITIONS: Type 2 Diabetes Mellitus; Overweight and Obesity
Keywords: Very low-calorie ketogenic diet; VLCKD; Type 2 diabetes; Overweight; Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Overweight; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Dietary Supplement: VLCKD — The analysis will focus on the observation of the evolution of anthropometric and clinical parameters,such as the improvement or normalization of HbA1c, as well as on the evolution of the hypoglycemic medication between patients who accept VLCKD method

SUMMARY:
There is a strong correlation between being overweight, specifically with abdominal fat, and type 2 diabetes mellitus (T2DM). Recent scientific literature has highlighted the connection between significant weight loss, specifically 15% or more of body weight, and its positive impact on body composition and glycemic profiles. In this study, the focus is on very low carbohydrate ketogenic diets (VLCKDs) as a nutritional strategy for managing excess weight and improving diabetes. Current research is transforming the understanding of T2DM, demonstrating that effective and timely interventions can lead to diabetes remission, including a partial recovery of insulin secretion and function.

However, the daily life of a diabetic patient in a clinical setting may not always mirror that of a patient participating in a study, who receives planned follow-up visits and close supervision. To address this discrepancy, this study aims to analyze a cohort of patient records with T2DM and overweight who have adopted a VLCKD, specifically through the PnK® Method, in a private diabetology practice. The goal is to assess the impact of VLCKD on glycemic control in real-life scenarios.

DETAILED DESCRIPTION:
The investigator wishes to carry out an observational, retrospective, uncontrolled, monocentric analysis on a group of patients with overweight and type 2 diabetes mellitus (T2DM).

The analysis will focus on the observation of the evolution of anthropometric and clinical parameters, such as the improvement or normalization of HbA1c, as well as on the evolution of the hypoglycemic medication.

The data collected and analyzed will correspond to 4 moments:

1. T0, at the start of treatment.
2. T1, at the end of VLCKD, period of ketosis with an average duration of 12 weeks.
3. T2, after 6-9 months of support and individualized therapeutic education for a new lifestyle.
4. T3, after 18-24 months of usual follow-up with 1 visit every 3 to 6 months.

The population included in the analysis consists of adults with T2DM, with a BMI greater than 25 kg/m2, followed in a diabetology office. This constitutes a form of selection of the population because people with more social, economic, linguistic difficulties, more complex pathologies will be better taken care of in a hospital environment.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of type 2 diabetes
* Being overweight (BMI > 25 kg/m^2) or obesity (BMI > 29.9 kg/m^2)
* Have wished to engage in a weight loss program according to the PnK® method
* Have accepted and signed the consent for the use of data

Exclusion Criteria:

* Pregnancy or lactation
* Type 1 diabetes
* Eating disorders
* Psychiatric disorders
* Have any contraindication for doing the active or ketogenic phase

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A patient cohort with overweight and type 2 diabetes.
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2023-01-30 (Actual); Primary Completion 2023-07-20 (Actual); Study Completion 2023-10-02 (Actual)

PRIMARY OUTCOMES:
Diabetes remission | 24 months
  Measured as HbA1c (%)

SECONDARY OUTCOMES:
Change in body weight | 24 months
  Measured as kilograms (kg)
Change in body fat | 24 months
  Measuared in percentage (%)
Change in visceral fat | 24 months
  Measuared in percentage (%)
Change in waist circumference | 24 months
  Measured in percentage (%)
Change in Body Mass Index (BMI) | 24 months
  Measured in kilogram per square meter (kg/m^2)
Number of type 2 diabetes remissions | 24 months
  Measured as count of participants
Decreases in poglycemic drug treatments | 24 months
  Measured as changes in the number of diabetes treatments

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Daniela Sofra, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided